CLINICAL TRIAL: NCT02804282
Title: Open Label Study to Evaluate Product Design Clinical Performance of a To-Be-Marketed Drug-Device Combination Product (sc2Wear Furosemide Combination Product) in Subjects With Chronic Heart Failure
Brief Title: Product Design Clinical Performance Study of sc2Wear Furosemide Combination Product
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-00001
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sc2Wear Furosemide Combination Product (Experimental): Drug-device combination product of buffered furosemide injection, (Furosemide Injection Solution), 8 mg/mL, and patch pump (sc2Wear Furosemide Pump) for subcutaneous administration of 80 mg dose delivered over 5 hours.
  Interventions: Combination Product: sc2Wear Furosemide

INTERVENTIONS:
Combination Product: sc2Wear Furosemide — Drug-device combination product of buffered furosemide injection, (Furosemide Injection Solution), 8 mg/mL, and patch pump (sc2Wear Furosemide Pump)

SUMMARY:
The proposed single-dose study aims to evaluate the product design clinical performance of the to-be-marketed drug-device combination product, the sc2Wear Furosemide Combination Product, in adult Subjects previously diagnosed with mild to advanced heart failure.

The study drug formulation is a buffered Furosemide Injection Solution, 8 mg/mL, (total dose equals 80 mg/mL) administered subcutaneously for a total of 5 hours. The study device is the sc2Wear Furosemide Pump adhered to the body using medical grade adhesive.

The objectives of this study are:

* To demonstrate that the to-be-marketed drug-device combination product performs as intended and delivers 80 mg of Furosemide subcutaneously in the abdominal area
* To assess safety and local tolerance of the drug-device combination product

DETAILED DESCRIPTION:
This study will be an open label, single-dose study to evaluate product design clinical performance of a to-be-marketed drug-device combination product (sc2WearTM Furosemide Combination Product) in up to 70 adult male and female Subjects previously diagnosed with mild to advanced heart failure (NYHA Class II-IV). The study was designed and powered to achieve "95/95" performance testing. Methodology: Each Subject will complete Screening, Treatment, and Follow-Up Phases on an outpatient basis. During the Screening Phase, all Subjects who sign the informed consent form and satisfy the inclusion/exclusion criteria will be enrolled into the trial. Drug administration may start on the day of enrollment or be scheduled within 3 days of completion of Screening assessments. However, if the treatment visit doesn't occur within 3 days of initial screening, subjects may be rescreened and treated within 3 days of rescreening. The Treatment Phase comprises a preprogrammed bi-phasic 5 hour drug administration. Treatment Day observations will commence with pre-placement assessments and continue until after device removal. Device preparation, placement and removal will be performed by study staff in accordance with product instructions of use. Removal will occur within 3 hours of completion of drug delivery (8 hours of start of administration). Subjects will return 5-7 days after the Treatment Day for a post treatment follow-up and photography.

Blood samples will be obtained for the measurement of plasma furosemide levels prior to start of the administration and once during the plateau phase (1-5 hours following activation). After preparation of the skin the device will be placed on the upper abdominal area by clinical study staff. Subjects are advised to avoid strenuous physical activity or activities that could expose the device to moisture such as swimming, bathing or showering. Participants will be informed that marked diuresis may ensue after activation, and that they should avoid travel, operating a vehicle or other situations without immediate access to bathroom facilities. For this study, up to 70 unique reusable components (Activator) will be used. Likewise, up to 70 single-use units (Cartridge) will be used. Following removal from the skin, the assembled device will be inspected and photographed by the site staff. The used device (assembled Cartridge and Activator) will be placed in a sealed container and returned for further inspection and measurement of residual volume in the device reservoir by a qualified laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Male and female Subjects ≥18 years of age
3. New York Heart Association (NYHA) Class II-IV Heart Failure.
4. In the opinion of the Investigator, able to participate in the study.
5. If Subject is on oral diuretic, willing to suspend the oral furosemide or other loop diuretic treatment on the day of treatment (use of oral diuretic within 8 hours of start of treatment is not permitted).
6. If Subject has significant body hair on the abdomen, willing to clip or shave the area where the device will be placed prior to treatment.
7. Has the ability to understand the requirements of the study, and is willing to comply with all study procedures.

Exclusion Criteria:

1. Contraindication to furosemide.
2. History of chronic skin conditions requiring medical therapy.
3. Skin reaction to medical adhesives or history of poor skin adherence of adhesives.
4. Any local abdominal skin condition on the day of treatment i.e. sunburn, rash, eczema, etc.
5. Diabetic patients currently using an insulin pump and/or interstitial glucose monitors.
6. Clinically significant abnormalities at Screening in safety laboratory tests.
7. Hypokalemia - Potassium of < 3.6 mmol/L.
8. Systolic BP (SBP) < 90 mm Hg.
9. Temperature > 38°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment.
10. History of major abdominal surgery affecting the site of device placement.
11. Participation in another trial, within 30 days prior to Screening.
12. History of hepatitis B, hepatitis C, or HIV
13. Evidence of current or recent alcohol abuse.
14. Female Subject who is pregnant or lactating.
15. Any surgical or medical condition that -in the opinion of the Investigator - may interfere with participation in the study or that may affect the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Absence of Major Product Failure | 1-5 hours
  Freedom from failures leading to infusion errors.

SECONDARY OUTCOMES:
Local Pain Tolerance | 1-5 hours
  Subject-reported pain using 11 point numeric rating scale of 0 to 10.
Local Skin Tolerance | 1-8 days
  Adhesive site skin inspection for erythema, edema and other local reactions using 8 point scale.
Incidence of treatment-emergent Adverse Events and Serious Adverse Events | 1-8 days

IPD SHARING:
Plan to Share IPD: No